CLINICAL TRIAL: NCT00636571
Title: Determining the Feasibility of Post-Operative Training for Patients Diagnosed With Non-Small Cell Lung Cancer
Brief Title: Feasibility of Exercise With Post-Op Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Lance Armstrong Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00005438
Record Dates: First submitted 2008-02-27; First posted 2008-03-14 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Exercise; Non-Small Cell Lung Cancer; Cardiopulmonary Fitness
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise — Upright bike intervention for post-surgical lung cancer survivors.

SUMMARY:
Primary Objective: To examine the effects of an exercise training program on cardiopulmonary fitness in early-stage postoperative non-small cell lung cancer patients undergoing adjuvant chemotherapy

Secondary Objectives:

Determine patients' adherence levels to such a program during adjuvant chemotherapy Explore the effects of exercise training on treatment compliance and toxicity, and quality of life.

To explore the effects of exercise training on markers of inflammation (e.g., c-reactive protein, immune response) in patients undergoing adjuvant chemotherapy for early-stage non-small cell lung cancer

DETAILED DESCRIPTION:
Using a single-group, prospective design, potential participants will be identified and screened for eligibility by the PI (LWJ) via medical record review of patients scheduled for their primary adjuvant chemotherapy consultation at DUMC and Durham VA. As a routine part of clinical care, during the treatment consultation the attending oncologist will perform a physical examination to screen for cardiovascular risk factors, the results of which will be recorded in the patients' medical records. Immediately following their consultation and oncologist approval, potential participants will be provided with a thorough review of the study by the principal investigator (LJ) and asked if they are willing to participate. Interested participants will be given an information package that provides further information on study participation. Two to five days following their treatment consultation and prior to the initiation of chemotherapy, interested participants will be contacted by telephone by the PI to answer any questions and to schedule the baseline assessment visit. At the baseline visit, participants will be asked to sign the informed consent and will be given a copy for their records. After consent, they will be given a baseline ECG and physician monitored cardiopulmonary exercise test (stress test) to screen for undiagnosed cardiovascular disease. Following the successful completion of baseline assessments, all participants will be scheduled for their initial exercise training session. Finally, on a different group of patients we will perform a random retrospective medical chart review of 50 completely-resected NSCLC patients who received usual care (i.e., no exercise training) during the study period to obtain comparative information on the treatment toxicity/compliance rate. The chart review will be performed by Drs. Jones, Garst and Crawford and will assess treatment toxicity and compliance over the entire course of adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Legal age (>18 years old)
* Absence of contraindications to chemotherapy
* Ability to read and understand English
* Signed informed consent prior to the initiation of study procedures
* Primary attending oncologist approval.

Exclusion Criteria:

* Acute myocardial infarction (3-5 days)
* Unstable angina
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
* Syncope
* Acute endocarditis
* Acute myocarditis or pericarditis
* Uncontrolled heart failure
* Acute pulmonary embolus or pulmonary infarction
* Thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Room air desaturation at rest ≤85%
* Respiratory failure
* Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
* Mental impairment leading to inability to cooperate.
* Finally, patients presenting with no medical history will not be eligible for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
ECG stress test | 8 weeks, 16 weeks

SECONDARY OUTCOMES:
Safety | 8 weeks, 16 weeks
adherence levels | 8 and 16 weeks
  The study will determine patients' adherence levels to such a program during adjuvant chemotherapy.
Treatment compliance and toxicity, and quality of life | 8 and 16 weeks
  The study will explore the effects of exercise training on treatment compliance and toxicity, and quality of life.
Inflammation | 8 and 16 weeks
  The study will explore the effects of exercise training on markers of inflammation (e.g., c-reactive protein, immune response) in patients undergoing adjuvant chemotherapy for early-stage non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jones, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States